CLINICAL TRIAL: NCT05709015
Title: Evaluation of a Mouthwash Formulation Containing Neutral Electrolysed Water on De-novo Plaque Formation, Gingival Inflammation, MMP-8 Activity and the Oral Microbiome
Brief Title: Plaque Inhibitory Effect of Neutral Electrolysed Water in the Form of a Mouthwash in a 4-day Non-brushing Model
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: EOWG
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-01

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis | interventions — chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 (Other): Based on a randomisation table, each participant will use either a mouthwash containing neutral electrolyzed water, placebo, or chlorhexidine digluconate twice a day instead of tooth brushing and flossing for 4 days. Each subject will receive each mouthwash type only once during the study period (he/she will receive a different mouthwash type in every arm of the study based on a randomisation table).
  Interventions: Other: Neutral electrolyzed water; Drug: Placebo; Drug: Chlorhexidine digluconate
- 2 (Other): Based on a randomisation table, each participant will use either a mouthwash containing neutral electrolyzed water, placebo, or chlorhexidine digluconate twice a day instead of tooth brushing and flossing for 4 days. Each subject will receive each mouthwash type only once during the study period (he/she will receive a different mouthwash type in every arm of the study based on a randomisation table).
  Interventions: Other: Neutral electrolyzed water; Drug: Placebo; Drug: Chlorhexidine digluconate
- 3 (Other): Based on a randomisation table, each participant will use either a mouthwash containing neutral electrolyzed water, placebo, or chlorhexidine digluconate twice a day instead of tooth brushing and flossing for 4 days. Each subject will receive each mouthwash type only once during the study period (he/she will receive a different mouthwash type in every arm of the study based on a randomisation table).
  Interventions: Other: Neutral electrolyzed water; Drug: Placebo; Drug: Chlorhexidine digluconate

INTERVENTIONS:
Other: Neutral electrolyzed water — Use of mouthwash containing neutral electrolyzed water twice daily for 4 consecutive days instead of tooth brushing and usage of interdental cleaning devices.
Drug: Placebo — Use of mouthwash containing placebo twice daily for 4 consecutive days instead of tooth brushing and usage of interdental cleaning devices.
Drug: Chlorhexidine digluconate — Use of mouthwash containing chlorhexidine digluconate twice daily for 4 consecutive days instead of tooth brushing and usage of interdental cleaning devices.

SUMMARY:
Electrolysed water (EOW) is produced by the electrolysis of sodium chloride in an aqueous solution, producing chlorine gas at the anode and sodium hydroxide and hydrogen at the cathode. EOW is known to have antimicrobial effects against various microorganisms, including viruses, bacteria, spores and fungi. Its antimicrobial activity is generally attributed to its hypochloric acid content - a product of chlorine gas dissolved in water. Due to its biocompatibility, known uses of EOW include ocular disinfection, nasal irrigation and chronic cutaneous wound care. In the dental setting, it may be used as a mouthwash, disinfectant, irrigant, mouthwash or dental gel.

The aim of this study is to investigate the effect of a mouthwash containing neutral electrolyzed water on plaque accumulation (evaluated using a disclosing agent and an intraoral scanner), gingival inflammation, MMP-8 activity and the oral microbiome. In this double-blind, cross-over, 4-day experimental gingivitis model, each subject will participate in all three arms of the study. Each arm will last 4 days, during which the subjects will be asked to refrain from toothbrushing and the use of interdental cleaning devices. Instead, they will be instructed to rinse their oral cavities twice daily with either EOW, placebo or a positive control (chlorhexidine), according to a randomisation chart (each subject will receive a different mouthwash type in every arm of the study). The outcomes will be assessed at baseline and after 4 days. A washout period of at least 7 days will be implemented between each study arm.

ELIGIBILITY:
Inclusion criteria:

* age 20 - 30 years,
* non-smoker,
* systemically healthy,
* without regular systemic medication,
* presence of at least 6 teeth in each jaw quadrant,
* plaque index < 10 % at baseline visit,
* absence of periodontal pockets measuring > 4 mm.

Exclusion criteria:

* known allergy or suspected hypersensitivity to chlorhexidine digluconate,
* gingivitis,
* regularly use of mouthwash as part of oral hygiene routine,
* antibiotic treatment in the last 6 months or during the observation period,
* pregnancy or lactation,
* fixed or removable prosthetic devices, dental implants.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
3D plaque score | baseline, 4 days
  Differences in plaque scores evaluated by optical scanning
Plaque index | baseline, 4 days
  Differences on plaque score evaluated using the Turesky Modification of the Quigley-Hein Plaque Index

SECONDARY OUTCOMES:
Modified Gingival Index | baseline, 4 days
  Differences in the gingival index evaluated using the Lobene Modified Gingival Index
Microbiologic profile of gingival crevicular fluid | baseline, 4 days
  To determine if the mouthwashes effect the presence of the most relevant periodontal pathogens (e. g. Aggregibacter actinomycetemcomitans) in gingival crevicular fluid
MMP-8 in gingival crevicular fluid | baseline, 4 days
  To determine if the mouthwashes effect the amount of MMP-8 in gingival crevicular fluid

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ljubljana, Ljubljana, Slovenia

REFERENCES:
- [Derived] Povsic K, Munjakovic H, Zayed N, Teughels W, Seme K, Fidler A, Gaspersic R. Electrolyzed saline as an alternative to chlorhexidine: Antimicrobial and biofilm volume outcomes in a 4-day non-brushing randomized controlled clinical trial. J Periodontol. 2026 Feb 2. doi: 10.1002/jper.70070. Online ahead of print. PMID 41627021